CLINICAL TRIAL: NCT03997890
Title: Clinical Outcomes of Patients Bilaterally Implanted With the TECNIS® Symfony or TECNIS® Symfony Toric Extended Range of Vision IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2016-0029
Record Dates: First submitted 2019-06-18; First posted 2019-06-25 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Cataract
Keywords: Extended depth of focus; Multifocal intraocular lens; Presbyopia; Cataract surgery
MeSH Terms: conditions — Cataract; Presbyopia | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Symfony group (Experimental): The subjects who underwent cataract surgery with binocular implantation of either Symfony or Symfony toric IOLs
  Interventions: Procedure: Cataract surgery with binocular implantation of either Symfony (ZXR00) or Symfony toric (ZXT) IOLs

INTERVENTIONS:
Procedure: Cataract surgery with binocular implantation of either Symfony (ZXR00) or Symfony toric (ZXT) IOLs — After creating an initial side port incision with a 15-degree blade, 3-step clear corneal incisions were made using a 2.5 mm disposable metal blade. Sodium hyaluronate 1.0% (Healon; Abbott Medical Optics) was then injected into the anterior chamber. A continuous curvilinear capsulorrhexis, measuring 5.5 mm in diameter, was generated using a 26 gauge bent needle. After hydrodissection, phacoemulsification was done to remove nuclear fragments and aspiration of residual cortex. In all eyes, a Symfony or Symfony toric IOL was implanted in the capsular bag using a disposable implantation system. Irrigation and aspiration were performed to minimize ophthalmic viscoelastic surgical device retention at the end of surgery. The main incision and side port were sealed with stromal hydration using a balanced salt solution.

SUMMARY:
In With increased patients' demand for a spectacle-free lifestyle and technological advancements, cataract surgery with multifocal intraocular lens (IOL) implantation has become an effective solution for correcting presbyopia in patients who want to maintain their full range of vision.

Conventional bifocal IOLs used either refractive or diffractive optics to split the light and create 2 principal focal points, thus providing functional vision at distance and near. This simultaneous imaging principle produces a sharp image that is overlaid by a secondary blurred out-of focus image, so these IOLs inherently produce a deterioration in contrast sensitivity and unwanted photic phenomena such as glare and halos. Additionally, studies reported insufficient intermediate vision with bifocal IOLs.

There is an increasing desire for spectacle independence at intermediate distance, especially due to the increased use of computers and smartphones. Trifocal IOLs were introduced to the market in 2010 and participants provide an additional, third focal point to improve intermediate vision without compromising distance and near vision. However, participants are still vulnerable to decreased contrast sensitivity and photic phenomena due to the IOL's mechanism of splitting the light into discrete focal points.

An extended depth of focus (EDOF) technology was recently introduced with the aim to improve intermediate vision while maintaining image contrast. The diffractive echelette design, embedded on its posterior optical surface, extends the range of vision and the achromatic technology reduces corneal chromatic aberrations to enhance retinal image quality and improve contrast sensitivity. The elongated focus allows imaging in a continuous range of vision without overlapping near and far images, and therefore theoretically would provide a more consistent distance and intermediate vision with less dysphotopsia.

The aim of this study was to investigate the clinical outcome of patients bilaterally implanted with either Tecnis Symfony or Tecnis Symfony toric extended range of vision IOLs (Johnson & Johnson Vision, Santa Ana, CA, USA) in terms of visual performance at different distances, spectacle independence, photic phenomena, and patient satisfaction.

DETAILED DESCRIPTION:
Enrollment period : 18 months after IRB approval Participants : Patients who had uncomplicated cataract surgery with binocular implantation of either Symfony (ZXR00) or Symfony toric (ZXT) IOLs.

Methods: The postoperative examinations were performed at 4-8 weeks, and 4-6 months postoperatively. Binocular corrected (CDVA) and uncorrected (UDVA) distance visual acuity was assessed at 4 m using a Snellen chart. Binocular uncorrected intermediate visual acuity (UIVA) at 70 cm and binocular uncorrected near visual acuity (UNVA) at 40 cm were assessed using the Rosenbaum near vision card.

A subjective questionnaire on spectacle use, photic phenomena, and satisfaction was administered to all patients. Patients were asked how often (never, occasionally, 50% of the time, frequently) participants wear spectacles for near, intermediate, and distance activities. Non-directed and directed questions were used with regard to visual symptoms. Photic phenomena (halos, glare and starbursts) were graded as none, trace, mild, moderate, or severe. Patients were asked to rate their level of satisfaction with distance, intermediate, and near vision on a scale from 0 (completely dissatisfied) to 10 (completely satisfied). Additionally, participants were asked whether participants would choose the same IOL again and if participants would recommend the IOL to their friends and family. Surgeons were also asked to rate their level of satisfaction on a scale from 0 to 10 in terms of the ease of manipulation and implantation of the IOL and the visual performance of the IOL.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of 20 years or older
* 2. Cataract

Exclusion Criteria:

* 1. Amblyopia
* 2. Keratoconus
* 3. Previous corneal or refractive surgery
* 4. Chronic or recurrent uveitis
* 5. Acute ocular disease
* 6. Previous ocular surgeries
* 7. Glaucoma
* 8. Any ocular disease which could possible affect the postoperative visual acuity

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Visual outcome | preoperative 4-6 weeks
  1. Uncorrected Distance Vision Acuity (4 meters) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 weeks
  2. Corrected Distance Vision Acuity (4 meters) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 weeks
  3. Uncorrected Intermediate Visual Acuity (70 cm) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 weeks
  4. Uncorrected Near Visual Acuity (40 cm) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 months
  1. Uncorrected Distance Vision Acuity (4 meters) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 months
  2. Corrected Distance Vision Acuity (4 meters) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 months
  3. Uncorrected Intermediate Visual Acuity (70 cm) in logMAR scale at each time point.
Visual outcome | preoperative 4-6 months
  4. Uncorrected Near Visual Acuity (40 cm) in logMAR scale at each time point.

SECONDARY OUTCOMES:
Spectacle use | Postoperative 4-6 weeks
  Patients were asked how often (never, occasionally, 50% of the time, frequently) participants wear spectacles for near, intermediate, and distance activities.
Spectacle use | Postoperative 4-6 months
  Patients were asked how often (never, occasionally, 50% of the time, frequently) participants wear spectacles for near, intermediate, and distance activities.
Photic phenomena | Postoperative 4-6 weeks
  Photic phenomena (halos, glare and starbursts) were graded as none, trace, mild, moderate, or severe.
Photic phenomena | Postoperative 4-6 months
  Photic phenomena (halos, glare and starbursts) were graded as none, trace, mild, moderate, or severe.
Patient Satisfaction | Postoperative 4-6 weeks
  Patients were asked to rate their level of satisfaction with distance, intermediate, and near vision on a scale from 0 (completely dissatisfied) to 10 (completely satisfied). Additionally, participants were asked whether participants would choose the same IOL again and if participants would recommend the IOL to their friends and family.
Patient Satisfaction | Postoperative 4-6 months
  Patients were asked to rate their level of satisfaction with distance, intermediate, and near vision on a scale from 0 (completely dissatisfied) to 10 (completely satisfied). Additionally, participants were asked whether participants would choose the same IOL again and if participants would recommend the IOL to their friends and family.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No